CLINICAL TRIAL: NCT03116009
Title: Randomization of Early Versus Standard Diabetes Screening Among Obese Pregnant Women
Brief Title: Randomization of Early Diabetes Screening Among Obese Pregnant Women.
Acronym: REDSOAP
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Former PI Left the Institution
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Mary Stephenson, Professor of Obstetrics and Gynecology, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-0737
Record Dates: First submitted 2017-02-08; First posted 2017-04-14 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Gestational Diabetes
Keywords: Obesity; Pregnancy; Diabetes Mellitus; Perinatal Outcomes
MeSH Terms: conditions — Diabetes, Gestational; Obesity; Diabetes Mellitus | interventions — Mass Screening; glutaminyl-peptide cyclotransferase; Glycated Hemoglobin

STUDY DESIGN:
Intervention Model Description: Two groups of obese pregnant women:
  Group 1: They will be screened for diabetes mellitus before 20 weeks of gestation.
  Group 2: They will be screened for diabetes mellitus at 24 - 28 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Screening for diabetes with 1-hour GCT and HbA1 (Active Comparator): Participants in this group will do 1-hour GCT before 20 weeks of gestation. Those with positive test will undergo 3-hours OGTT. Diabetes will be diagnosed if they have two or more abnormal values out of the 4 values and they will be treated accordingly based on the institutional protocol. They will also have HbA1C done.
  Interventions: Drug: Screening for diabetes with 1-hour GCT and HbA1
- Early screening with only HbA1C (Experimental): Participants in this group will only have HbA1C done before 20 weeks but will do the standard diabetes screening at 24 - 28 weeks. Those who have abnormal values will also be treated based on the institutional protocol.
  Interventions: Drug: Screening for diabetes with 1-hour GCT and HbA1

INTERVENTIONS:
Drug: Screening for diabetes with 1-hour GCT and HbA1 — They will receive 50gm oral glucose tolerance test before 20 weeks and if abnormal, they will do the diagnostic test with 100gm OGTT with HbA1C.
  Other Names: Early screening with only HbA1C

SUMMARY:
This will be a randomization of two groups of obese pregnant women into early screening for diabetes mellitus at the time of their first or subsequent prenatal visits before 20 weeks of gestation versus standard time of screening for diabetes at 24 - 28 weeks as it is done for all pregnant women. The perinatal outcomes between the two groups will be compared to determine whether early screening for diabetes in all obese pregnant women has a clinical merit or significant.

DETAILED DESCRIPTION:
As part of normal physiological changes of pregnancy, there is increased insulin resistance, which causes dysregulation of maternal glucose homeostasis. Obesity, which is body mass index greater or equal to 30 kg/m2, is also associated with impaired glucose metabolism. Women with higher body mass index (BMI) usually have higher risk of developing gestational diabetes mellitus (GDM) than normal BMI women. The American Congress of Obstetricians and Gynecologists (ACOG) recommends early screening for gestational diabetes mellitus in certain categories of patients with higher risk factors which includes previous medical history of gestational diabetes mellitus, known impaired glucose metabolism and obesity.

However, there is poor compliance by many clinicians of this ACOG recommendation.. One of the reasons for the poor compliance is that it was based on expert opinion and consensus which is level III evidence. There has not been any robust study to determine the clinical importance of screening obese women early versus screening them at the same time like every pregnant women at 24 - 28 weeks.

The justifications for recommendation for early diabetes screening are:

1. It will help diagnose pre-existing type 2 DM unrecognized prior to pregnancy. Uncontrolled pre-gestational type 2 DM in the first trimester has been shown to have the same maternal and perinatal adverse effects as type 1 DM.
2. It will help detect women with impaired glucose metabolism, in which early interventions may prevent the development of GDM later on in pregnancy and its associated complications.
3. Treatment of type 2 diabetes in the first trimester will minimize adverse maternal and perinatal outcomes such as congenital malformation, hypertension or preeclampsia often associated with poorly controlled diabetes.

However, there is currently no strong evidence to support that early GDM screening in obese pregnant women is cost effective or is beneficial in reducing maternal and perinatal adverse outcomes despites its recommendation by many professional societies.

Objectives of this study:

1. Primary objectives:

   1. To compare the rate of neonatal large for gestational age (> 90 percentile) or macrosomia (> 4000gm birth weight) between the two groups: The study group and the control group.
   2. To compare the rate of neonatal large for gestational age (> 90 percentile) or macrosomia (> 4000gm) between participants with diabetes diagnosed at early screening and those with true gestational diabetes diagnosed at 24 - 28 weeks. Those with true GDM are those who test negative during early screening but become positive at 24 - 28 weeks of gestation.
2. Secondary objectives:

   1. To compare pregnancy outcomes between the early screening group and the control group. Maternal outcomes will include the development of pre-eclampsia, pregnancy induced hypertension, maternal weight gain during pregnancy, and 3rd or 4th degree perineal lacerations. Perinatal outcomes will include rate of miscarriage, preterm delivery, intra-uterine growth restriction, intra-uterine fetal death and neonatal metabolic complications (hypoglycemia, hypocalcaemia or hyperbilirubinemia).
   2. To compare pregnancy outcomes between diabetes diagnosed at early screening and true gestational diabetes diagnosed at 24 - 28 weeks.
   3. To describe characteristics of participants in each group including medical co-morbidities and obstetric complications.
   4. To determine glycemic control by measurement of HbA1C at the time of diagnosis of diabetes and at term, prior to delivery.
   5. To compare composite neonatal complications between the two groups such as NICU admission, duration of NICU stay, respiratory distress syndrome, neonatal sepsis, necrotizing enterocolitis, intra-ventricular hemorrhage and neonatal death.
   6. To determine sensitivity and specificity of early diabetes screening across the obesity classes according to the world health organization (WHO) classification.
   7. Cost analysis of early diabetes screening among obese pregnant women. The duration of this study will be approximately 2 years; obese pregnant women will be enrolled September 2016 to August 2017, and they will be followed to the end of their pregnancy.

      * This will be a randomized controlled trial of two groups of obese pregnant women. The study group will receive early diabetes screening (a GCT) during their first prenatal clinic visit or a subsequent visit at less than 20 weeks of gestation. The control group will be screened at 24 - 28 weeks of gestation, which is the time all low risk pregnant women are screened.
      * The study will be performed in the Center for Women's Health and Mile Square health center of the University of Illinois Hospital and Health Science System (UI Health). The providing physician, midwife or trained recruiters will recruit participants from these two sites if they meet eligibility criteria.
      * Eligible participants will be approached and counseled about the nature of the study. If they are willing to participate, informed consent would be obtained from them and a questionnaire to obtain vital clinical information would be administered. Thereafter, they would be instructed to go to the laboratory to perform 1 hour 50 g glucose challenge test (GCT) with HbA1C (study group) or HbA1C only (control group). The 1-hour GCT involves administration of 50g of glucose solution by mouth. Participants do not need to be fasting. After 1 hour, venous blood will be drawn along with other prenatal labs, and glucose level and HbA1C would be analyzed. The control group will not be given the 1-hour GCT but only perform HbA1C level during their routine prenatal lab tests. Practitioners at UIC routinely request the HbA1C test as standard of care for obese pregnant women at early gestation based on ACOG recommendation.
      * As part of standard clinical care, if a pregnant patient has a positive 1-hour GCT at any point in her pregnancy (defined by plasma glucose level of 140 mg/dl or greater) they are to receive a 3-hour 100g oral glucose tolerance test (OGTT) at a later date. In this test, the patients are advised to avoid smoking or alcohol for 3 days preceding the test date, although they may continue with their regular diet during this period. The patient is instructed to fast over-night for 8 -10 hours prior to the test. A 2.5 ml blood sample is drawn for the fasting plasma glucose level, then a 100 g glucose solution is given to the patient orally. A 2.5 ml blood sample is then drawn each at 1, 2 and 3 hours. A diagnosis of diabetes mellitus is made if there are two or more abnormal plasma glucose values using the Carpenter and Coustan criteria (Fasting plasma glucose > 90 mg/dl, 1 hour > 180 mg/dl, 2 hours > 155 mg/dl and 3 hours > 140 mg/dl) 21. A random plasma glucose or 1-hour 50 g GCT> 200 mg/dl will also be considered as diagnostic of diabetes mellitus and will no require the 3-hours OGTT.
      * As part of standard clinical care, those diagnosed with DM would receive diabetic teaching and would be referred to a dietitian for nutritional counseling. Patients would be taught on how to monitor daily blood glucose at home and come back 1 - 2 weeks later for evaluation where they would be evaluated for glycemic control. If the blood glucose values are within normal range, patient would continue with dietary intervention only. However, if the blood glucose values are abnormal, they would be given oral hypoglycemic drugs (Metformin or Glyburide), or insulin according to the discretion of the provider. All pregnant diabetic patients on medications are usually managed in the high risk OB clinic at UIC.
      * Those in the study group that test negative to the 1-hour GCT and 3-hour OGTT, and the participants in the control group will be followed routinely according to their medical and / or other obstetric conditions. At 24 - 28 weeks, they will undergo a 1-hour GCT and those that test positive will be also have the 3-hour OGTT based on current ACOG recommendation. If they are diagnosed with diabetes, they would receive the same standard-of-care interventions or treatments as necessary.

Note: those patients in the early screening group who have a negative GCT or OGTT at the < 20week prenatal visit will not be charged for the GCT at the 24-28week visit.

* As part of standard clinical care, participants will be followed until delivery in a manner appropriate to their clinical or other medical and obstetric conditions. Data would be collected via the administered questionnaire and also from the participants' electronic medical records. Additionally, the records of the participant's newborns will be reviewed in order to collect neonate outcomes.
* The questionnaire will be used to collect baseline data such as medical record number, maternal age, race / ethnicity, educational level, employment status, nature of job, BMI, gravidity, parity, social and family history, obstetric history, medical and surgical history, and medications.

ELIGIBILITY:
Inclusion Criteria:

1. Obese pregnant women with BMI > 30 kg/m2
2. First prenatal visit or subsequent visit prior to 20 weeks of gestation
3. Maternal age > 18 years
4. Willingness to participate in the study and give informed consent

Exclusion Criteria:

1. Pre-existing DM or pre-gestational diabetes mellitus,
2. Gestational age more than 20 weeks at time of enrollment
3. Unknown or inability to determine gestational age even with last menstrual period
4. Previous medical history of gestational diabetes mellitus.
5. Known impaired glucose metabolism
6. HbA1C > 6.5 %

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only obese pregnant women
Enrollment: 600 (Actual)
Dates: Start 2017-03-19 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Large for gestational age or macrosomia | To be assessed within 2 days after delivery.
  Birth weight of newborn more than 90 percentile or birth weight of 4000gm or more will be assessed at the completion of that pregnancy.

SECONDARY OUTCOMES:
Maternal medical complications | For 6 months during antepartum and 6 weeks postpartum.
  Development of preeclampsia
Birth injuries | To be assessed within 2 days of delivery.
  Third or 4th degree perineal lacerations will be assessed soon after successful vaginal delivery either spontaneous or with assisted vaginal delivery.
Mode of delivery | To be assessed within 2 days of delivery.
  Normal vaginal delivery, operative vaginal delivery or cesarean section
Glycemic control | To be assessed during pregnancy and 6 weeks postpartum.
  Use of HbA1C, and postpartum glucose challenge test as postpartum visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mary D Stephenson, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No